CLINICAL TRIAL: NCT06477705
Title: Energy Expenditure Induced by Football Training in Overweight Middle-aged Males
Brief Title: The Energy Cost of 1-Hour Football Training
Acronym: FAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FAM_EE
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Energy Expenditure; Body Composition; Resting Metabolic Rate; Overweight and Obesity
Keywords: Football training; Energy Expenditure; Oxygen consumption; Blood lactate; Metabolic Syndrome
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in this arm will receive no intervention
- Recreational Football Training (Experimental): Participants in this arm will participate in a football training session for 60 minutes. During the training the participans will execute the warm-up process, the part of soccer technical exercises and they will play a small-side-game.
  Interventions: Other: FAM

INTERVENTIONS:
Other: FAM — Participants will perform a recreational Football Training session for 60 minutes. The training will include the warm-up, soccer technical exercises and a small-side game
  Arms: Recreational Football Training

SUMMARY:
This study aims at investigating the energy expenditure following a single Football trainning session in middle aged males. The participants will perform a soccer training session [A single training session including 60 minutes of warm up, soccer technical exercises and small-sided game] and a cotrol trial (No intervention included, only daily measurements) in randomized, repeated measures, crossover design.

DETAILED DESCRIPTION:
Football is an intermittent sport with frequent activity changes and a high number of explosive movements. As a result, both mitochondrial and the non-mitochondrial energy sources (phosphagens, lactic acid system) are heavily utilized during football practice and games, which may contribute to the rise of oxygen consumption following exercise (EPOC) compared with cardiovascular-type exercise, where VO2 can reach a steady state.However, it is observed that there is a methodological limitation in the determination of total energy expenditure during and after football training and specifically in overwight middle-aged participans with metabolic syndrome.

Twenty overweight middle-aged males with mtabolic syndrome will perform a soccer training session [A single training session including 60 minutes of warm up, soccer technical exercises and small-sided game] and a cotrol trial (No intervention included, only daily measurements) in randomized, repeated measures, crossover design. Anthropometric, biochmeistry indicators, metabolic, blood pressure, physical activity and performance measurements will be measured at baseline. Global positoning system and accelerometry devices will be used to measure the distance and intensity of football trianing. The metabolic cost will be estimated from heart rate, blood lactate, resting oxygen uptake, exercise oxygen uptake, and excess post-exercise oxygen consumption measurements using a portable gas analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Free of musculoskeletal injuries
* No use of ergogenic supplements or medication
* Free of chronic diseases
* age of 40-60 years
* BMI>25
* Metabolic syndrome

Exclusion Criteria:

* Musculoskeletal injury
* Use of alcohol, caffeine and any type of ergogenic supplements or medication during the course of the study

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-23 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-07-08 (Estimated)

PRIMARY OUTCOMES:
Change in exercise-induced energy expenditure | At pre-exercise, during, and post-exercise session (single bout lasting 60 minutes)
  Exercise energy expenditure (kcal) will be measured using a portable indirect calorimetry system
Change in excess post-exercise oxygen consumption (EPOC) | At post-exercise session (single bout lasting 60 minutes)
  EPOC (kcal) will be measured using a portable indirect calorimetry system
Change in blood lactate concentration (BLa) | At pre- and post-exercise session (single bout) at 3 minutes post-exercise
  BLa (mmol/L) concentration will be measured in a microphotometer with commercially available kits.
Change in heart rate | At pre-exercise, during, and post-exercise session (single bout lasting 60 minutes)
  Heart rate (bpm) will be measured with a wearable heart rate monitor
Change in perceived exertion | At pre-exercise and post-exercise session (single bout lasting 60 minutes)
  Rating of perceived exertion (RPE) will be measured with the Borg scale (0-10)
Respiratory Exchange Ratio (RER) | At pre-exercise, during, and post-exercise session (single bout lasting 60 minutes)
  Respiratory Exchange Ratio (RER) will be measured using a portable indirect calorimetry system
Breath Frequency (BF) | At pre-exercise, during, and post-exercise session (single bout lasting 60 minutes)
  Breath Frequency (BF) will be measured using a portable indirect calorimetry system

SECONDARY OUTCOMES:
Body weight | At baseline
  Body weight will be measured on a beam balance with stadiometer
Body height | At baseline
  Body height will be measured on a beam balance with stadiometer
Body mass index (BMI) | At baseline
  BMI will be calculated using the Quetelet's equation
Waist circumference (WC) | At baseline
  WC (cm) will be measured using a Gullick II tape
Hip circumference (HC) | At baseline
  HC (cm) will be measured using a Gullick II tape
Waist-to-hip ratio (WHR) | At baseline
  WHR will be calculated by dividing the waist by the hip measurement
Resting metabolic rate (RMR) | At baseline
  RMR (kcal) will be measured using a portable open-circuit indirect calorimeter with a ventilated hood system
Body fat (BF) | At baseline
  Body fat (%) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat mass (FM) | At baseline
  FM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Fat-free mass (FFM) | At baseline
  FFM (kg) will be assessed by whole-body dual-energy X-ray absorptiometry (DXA)
Bone mass density | At baseline
  Bone mass density will be measured by using Dual-emission X-ray absorptiometry
Bone mass content | At baseline
  Bone mass content will be measured by using Dual-emission X-ray absorptiometry
Peak Maximal oxygen consumption (Peak VO2) | At baseline
  Peak VO2 will be estimated by open circuit spirometry via breath by breath method
Dietary intake | At baseline
  Dietary intake will be assesed over a 7-day period using diet recalls
Field activity during the soccer training | [Time Frame: During the 60 minutes soccer training (ST) session (72 hours after baseline measurements)
  The field activity will be continuously monitored during the soccer training using global positioning system (GPS)
Systolic Blood Pressure | At baseline
  Systolic Blood Pressure will be examined using sphygmomanometer
Dystolic Blood Pressure | At baseline
  Dystolic Blood Pressure will be examined using sphygmomanometer
Rest Heart Rate | At baseline
  The rest heart rate will be estimated using a heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, Principal Investigator — University of Thessaly
Locations (1):
- Laboratory of Exercise Physiology, Exercise Biochemistry and Sports Nutrition, School of Physical Education, Sports Sciences and Dietetics, University of Thessaly, Trikala, Greece